CLINICAL TRIAL: NCT00105040
Title: A 19-week, Randomized, Double-blind, Multicenter, Placebo-controlled Safety Study to Evaluate the Cognitive and Neuropsychological Effects of Levetiracetam 20 - 60 mg/kg/Day, Divided in Twice Daily Dosing, as Adjunctive Treatment in Children 4 - 16 Years Old, Inclusive, With Refractory Partial Onset Seizures
Brief Title: A 19-week Cognition Study of Levetiracetam in Children With Partial Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N01103; 2014-004396-23 (EudraCT Number)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Epilepsy, Partial
Keywords: Partial onset seizures; epilepsy; levetiracetam; Keppra; cognition; behavior; pediatry
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Behavior | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (LEV) (Experimental): Oral tablets or oral solution at 20-60 mg/kg/d, divided into twice daily dosing.
  Interventions: Drug: Levetiracetam
- Matching Placebo (PBO) (Placebo Comparator): Oral tablets and oral solution.
  Interventions: Other: Placebo (PB)

INTERVENTIONS:
Drug: Levetiracetam — Oral tablets or oral solution at 20-60 mg/kg/d, divided into twice daily dosing.
  Other Names: Keppra
  Arms: Levetiracetam (LEV)
Other: Placebo (PB) — Oral tablets and oral solution
  Arms: Matching Placebo (PBO)

SUMMARY:
A 12-week Evaluation Period will be used to characterize potential cognitive and neuropsychological effects of LEV (20 - 60 mg/kg/day), as adjunctive treatment in children 4 - 16 years old, inclusive, with refractory partial onset seizures when compared to adjunctive treatment with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects (4 - 16 years old) diagnosed with refractory partial onset seizures for a minimum of six months prior to Visit 1 experiencing at least two partial onset seizures during the four weeks prior to Visit 1 will be enrolled
* Subjects should be on a stable regimen of one or a maximum of two other antiepileptic drugs (AEDs) for at least 2 weeks prior to Visit 1
* Subject must have an Intelligence Quotient (IQ) as assessed during Visit 1 of at least 70
* Subject and parent/guardian should be fluent in English

Exclusion Criteria:

* Subject must not have had previous treatment with levetiracetam unless, in the opinion of the investigator, the subject's previous treatment was inadequate in dose or duration to provide an accurate assessment of the therapy, or the effect of levetiracetam was confounded by concomitant medication
* Subject is receiving benzodiazepines on a routine or chronic basic and is unable to discontinue use four weeks prior to Visit 1
* Subject has seizures too close together to accurately count
* Subject has a current psychiatric disorder other than mild to moderate attention deficit, behavior, or learning disorders

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2004-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Leiter International Performance Scale-Revised (Leiter-R) Attention and Memory (AM) Battery's Memory Screen Composite Score from Baseline (Visit 2) to the end of the Evaluation Period (Week 12 or Early Discontinuation Visit) | Baseline (Visit 2) to the end of the Evaluation Period (Week 12 or Early Discontinuation Visit)
  The Leiter-R includes two groupings of sub-tests: (1) the Visualization and Reasoning (VR) Battery with 10 sub-tests of nonverbal intellectual ability related to visualization, reasoning, and spatial ability; and (2) the Attention and Memory (AM) Battery with 10 sub-tests of nonverbal attention and memory function. The Examiner Rating Scale has 49 items that describe the child's activity level, attention, impulse control, and other emotional characteristics that may interact with test performance. The focus of the items is on actions, verbalizations, moods and other behaviors of the child. The examiner rates the child using the following scale: 0 = rarely or never; 1 = sometimes; 2 = often; 3 = usually or always.

SECONDARY OUTCOMES:
Change from Baseline in Wide Range Assessment of Memory and Learning-Second Edition (WRAML-2) General Memory from Baseline to Week 12 or Early Discontinuation Visit (EDV) | Baseline to Week 12 or EDV
  The WRAML-2 is comprised of 2 Verbal, 2 Visual, and 2 Attention-Concentration sub-tests, yielding a Verbal Memory Index, a Visual Memory Index and an Attention-Concentration Index. Together these sub-tests yield a General Memory Index. Scaled and standard scores allow performance comparisons based on age and 4 delayed recall sub-tests include guidelines for determining the level of recall. A composite General Memory Index score will be computed.
Change from Baseline in Wide Range Assessment of Memory and Learning-Second Edition (WRAML-2) Visual Memory Index from Baseline to Week 12 or Early Discontinuation Visit (EDV) | Baseline to Week 12 or EDV
  The WRAML-2 is comprised of 2 Verbal, 2 Visual, and 2 Attention-Concentration sub-tests, yielding a Verbal Memory Index, a Visual Memory Index and an Attention-Concentration Index. Together these sub-tests yield a General Memory Index. Scaled and standard scores allow performance comparisons based on age and 4 delayed recall sub-tests include guidelines for determining the level of recall. A composite General Memory Index score will be computed.
Change from Baseline in Wide Range Assessment of Memory and Learning-Second Edition (WRAML-2) Verbal Memory Index from Baseline to Week 12 or Early Discontinuation Visit (EDV) | Baseline to Week 12 or EDV
  The WRAML-2 is comprised of 2 Verbal, 2 Visual, and 2 Attention-Concentration sub-tests, yielding a Verbal Memory Index, a Visual Memory Index and an Attention-Concentration Index. Together these sub-tests yield a General Memory Index. Scaled and standard scores allow performance comparisons based on age and 4 delayed recall sub-tests include guidelines for determining the level of recall. A composite General Memory Index score will be computed.
Change from Baseline in Wide Range Assessment of Memory and Learning-Second Edition (WRAML-2) Attention/Concentration Index from Baseline to Week 12 or Early Discontinuation Visit (EDV) | Baseline to Week 12 or EDV
  The WRAML-2 is comprised of 2 Verbal, 2 Visual, and 2 Attention-Concentration sub-tests, yielding a Verbal Memory Index, a Visual Memory Index and an Attention-Concentration Index. Together these sub-tests yield a General Memory Index. Scaled and standard scores allow performance comparisons based on age and 4 delayed recall sub-tests include guidelines for determining the level of recall. A composite General Memory Index score will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (45):
- United States (38):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Los Angeles, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Gainesville, Florida
  - Loxahatchee Groves, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Voorhees Township, New Jersey
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Germantown, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Galveston, Texas
  - Houston, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Canada (3):
  - Scarborough Village, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
- South Africa (4):
  - Bloemfontein
  - Cape Town
  - Capitol Park
  - Johannesburg

REFERENCES:
- [Result] Levisohn PM, Mintz M, Hunter SJ, Yang H, Jones J; N01103 Levetiracetam Study Group. Neurocognitive effects of adjunctive levetiracetam in children with partial-onset seizures: a randomized, double-blind, placebo-controlled, noninferiority trial. Epilepsia. 2009 Nov;50(11):2377-89. doi: 10.1111/j.1528-1167.2009.02197.x. Epub 2009 Aug 21. PMID 19702752
- [Result] de la Loge C, Hunter SJ, Schiemann J, Yang H. Assessment of behavioral and emotional functioning using standardized instruments in children and adolescents with partial-onset seizures treated with adjunctive levetiracetam in a randomized, placebo-controlled trial. Epilepsy Behav. 2010 Jul;18(3):291-8. doi: 10.1016/j.yebeh.2010.04.017. Epub 2010 May 23. PMID 20547106